## **Informed Consent Form**

<u>Title</u>: Inflammation-Induced CNS Glutamate Changes in Depression

NCT Number: NCT03004443

Version Date: October 23, 2019

## You Are Being Asked to Be in a Research Study

## What Is a Research Study?

The main purpose of research studies is to gain knowledge. This knowledge may be used to help others. Research studies are not intended to benefit you directly, though some might.

## **Do I Have to Do This?**

No. Being in this study is entirely your choice. If you decide to join this study, you can change your mind later on and withdraw from the research study.

Taking part in a study is separate from medical care. The decision to join or not join the research study will not affect your status as a patient.

## What Is This Document?

This form is an informed consent document. It will describe the study risks, procedures, and any costs to you.

This form is also a HIPAA Authorization document. It will describe how your health information will be used and by whom.

Signing this form indicates you are willing to take part in the study and allow your health information to be used.

## What Should I Do Next?

- 1. Read this form, or have it read to you.
- 2. Make sure the study doctor or study staff explains the study to you.
- 3. Ask questions (e.g., time commitment, unfamiliar words, specific procedures, etc.)
- 4. If there will be medical treatment, know which parts are research and which are standard care.
- 5. Take time to consider this, and talk about it with your family and friends.

Document Approved On: «ApproveDate»

# Emory University Consent to be a Research Subject / HIPAA Authorization

<u>Title</u>: Inflammation-Induced CNS Glutamate Changes in Depression

Principal Investigator: Andrew H. Miller MD and Ebrahim Haroon MD

**Sponsor:** National Institute of Mental Health (NIMH)

## Introduction

You are being asked to be in a medical research study. This form is designed to tell you everything you need to think about before you decide if you want to be a part of the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study. The decision to join or not join the research study will not cause you to lose any medical benefits. If you decide not to take part in this study, your doctor will continue to treat you.

## Before making your decision:

- Please carefully read this form or have it read to you
- Please listen to the study doctor or study staff explain the study to you
- Please ask questions about anything that is not clear

You can take a copy of this consent form, to keep. Feel free to take your time thinking about whether you would like to participate. You may wish to discuss your decision with family or friends. Do not sign this consent form unless you have had a chance to ask questions and get answers that make sense to you. By signing this form you will not give up any legal rights.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. law. This Web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time.

## What is the purpose of this study?

You are being asked to volunteer for a research study because you have been diagnosed with major depression. The purpose of this study is to understand how increased inflammation, a process called immune activation, causes a change to our normal brain chemistry to fuel symptoms of depression. Also, this study will determine whether a medicine called infliximab will improve symptoms of depression by decreasing inflammation. Infliximab is also known by its brand name Remicade. Infliximab (Remicade), is given to people by an IV needle. It is currently used to treat two illnesses: rheumatoid arthritis and Crohn's disease. Infliximab is thought to help these conditions because it reduces inflammation in the body. For this reason, researchers think that a drug like infliximab, which reduces inflammation, may be helpful in treating symptoms of depression in people with high inflammation. Still, it is important to point out that the Food and Drug Administration has not approved infliximab for treating depression. It is possible that the researchers will learn something new during the study about the risks of being in it. If this happens, they will tell you about it. Then you can decide if you want to continue to be in this study or not. You may be asked to sign a new consent form that includes the new information if you decide to stay in the study.

Before you agree to take part in this study, please read this consent form and ask as many questions as you need to be sure you understand the possible risks and benefits. You may talk to family and friends about your decision. Please take your time to make your decision. Should you decide to participate in this study, you are free to change your mind at any time without penalty or loss of any benefit.

 Version Date: 10/23/2019

IRB Form 04152016

Document Approved On: «ApproveDate»

This consent form contains important facts to help you decide if it is in your best interest to take part in this study. If you have any questions that are not answered in this consent form, one of the research staff will be happy to give you further information.

Two hundred male and female participants with depression, between the ages of 21-65 years, will be enrolled into the study. Sixty participants will be randomized to study medication or placebo. Your participation, should you decide to enter the study, will last about a month, including your screening visit(s).

Before you can participate in this study, you will need to come in for a screening visit to see if you are eligible to enter the study. The investigator and/or the investigator's staff will ask you questions and run tests that are described below to determine if you are eligible to enter the study. It is important that you answer all of the questions honestly and completely. If your condition or circumstances change during the study, you must tell the investigator.

If you are currently doing well on antidepressant medication, you will not be eligible to participate in this study. It would not be in your best interest to discontinue medication that is helping you. On the other hand, you may enter this study if you are not currently taking an antidepressant, mood stabilizer or any other psychotropic medication.

If you plan to take any medication or undergo any medical treatment other than taking the study infusion given to you, please notify the study team before starting the medication or treatment. This includes medications given to you or recommended by any other doctor, and over-the-counter drugs such as cough treatments, cold treatments, pain medications such as aspirin or ibuprofen, investigational drugs/procedures and sleeping medications. If elective surgery or a diagnostic procedure is planned the investigator has to be notified before the procedure is performed.

## **Medications to Avoid:**

You will be excluded from the study if you take any of the following medications on a regular basis or if they are prescribed by a physician: psychiatric medication (for example: antidepressants, mood stabilizers, etc.) aspirin or aspirin-like compounds, ibuprofen or naproxen (for example: Advil, Aleve, Motrin IB), cholesterol medications (for example: simvastatin, Lipitor, Pravachol), antibiotics, topical steroids (i.e. hydrocortisone), vaccinations, herbal medications and omega-3 supplements. Please contact us if your doctor prescribes any new medication while participating in the study. Please also contact us if you plan on starting any new over-the-counter medications between study visits. Please do not stop taking any prescribed medications. If you take above medications on an as-needed (prn) basis, we will determine your eligibility to participate in the study based on frequency and necessity of intake and may need to discuss this with the prescribing physician before arriving at this decision

Although it is recommended that you do not drink alcoholic beverages during your participation in the study, you may drink alcohol on occasion (at most 1 glass of wine or equivalent per day). Use of illegal drugs during your participation in the study is not allowed and you will be drug-tested for illegal drugs as part of this study.

If the study doctor (Dr. Miller or his designee) determines that your depression has gotten worse at any time during the study, you may be discontinued from the study. When you have completed or been discontinued from the study, the study doctor will discuss how to best continue your treatment for depression. In addition, the study team will try to find a physician for follow up care if you do not have one.

During this study you will interact with study doctors, research clinicians and nurses trained to infuse infliximab. You will also interact with a research coordinator and other staff who will help arrange your schedule during the study.


## **Study Procedures:**

If you agree to participate, this is what will happen during the study. You will be screened first to see if you are a good match for the study. If you qualify, **the study visits will be spread across ~ 4 weeks.** 

**Table 1. Schedule of Study Procedures and Assessments** 

| Assessments | Intake | Screening | Base | Baseline* | | Day 3 | Week 1 | Week 2 | | 30 Day |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Visit | Visi | | | | Visit 1 | Visit 2 | F/U |
| | | | 1 | t 2 | | | | | | Phone |
| | | | | | | | | | | Call |
| Intake forms and assessments: Consent, HIPPA tracking, Release of Information**, | | | | | | | | | | |
| Consent of Means of Communication**, | | | | | | | | | | |
| Participant Payment Form**, MRI Screening | v | | | | | | | | | |
| Form**, Patient Health Questionnaire (PHQ-9)** or Clinician-Assisted QIDS-16 SR **, | Х | | | | | | | | | |
| Medication Avoidance List**, Lumbar Puncture | | | | | | | | | | |
| Information Guide, Schedule Quick Guide | | | | | | | | | | |
| Psychiatric screening: WRAT-3**, MMSE**, | | | | | | | | | | |
| HAM-D**, ATRQ, SCID V**, CSSRS, Clinical | | | | | | | | | | |
| Interview Review [to be done in place of imported | | X | | | | | | | | |
| psych assessments from prior study] | | | | | | | | | | |
| Laboratory Screening: Anti-nuclear AB**, C- | | | | | | | | | | |
| reactive protein, TSH, Hepatitis B surface | | | | | | | | | | |
| antigen**, Hepatitis C antibody**, HIV | | х | | | | | | | | |
| antigen/antibody**, QuantiFERON-TB Gold or | | ^ | | | | | | | | |
| TB Gold Plus, Rapid CRP Finger Prick [if | | | | | | | | | | |
| necessary to verify CRP], EKG, CXR | | | | | | | | | | |
| Serum pregnancy test | | Х | | Х | | | | Х | | |
| Medical History and Physical Examination or | | x | х | | [X] | х | [X] | x | [X] | |
| medical update | | | | | L-3 | | F-3 | | L-3 | |
| Adverse events, Concomitant medications | | | | | | ., | | | | |
| [Con. Med. not completed at 30 day F/U phone call | | X | Х | Х | [X] | Х | [X] | X | [X] | Х |
| only] | | | - | | | | | | | |
| Vital Signs, weight, height [screen only], waist- | | Х | х | Х | [X] | х | [X] | х | [X] | |
| hip ratio [screen only] Routine Labs: CBC with differential, urinalysis | | | | | | | | | | |
| w/ micro, comprehensive metabolic panel <sup>0</sup> | | Х | | Х | | | [X] | Х | [X] | |
| Urine toxicology | | Х | Х | Х | [X] | Х | [X] | Х | [X] | |
| Psychiatric baseline: Demographic Data**, | | | | | [A] | | [7] | | [7] | |
| CTQ**, Bipolarity Index** | | | Х | | | | | | | |
| Infusion (Infliximab or placebo) | | | | Х | | | | | | |
| Estrogen/progesterone | | | | Х | | | | | | |
| Urine pregnancy test | | | Х | | | Х | Х | Х | | |
| Research blood: Cytokine Multiplex, mRNA, | | | | v | [V] | v | [V] | v | | |
| Plasma CRP | | | Х | Х | [X] | X | [X] | Х | | |
| Clinician-Administered: SHAPS-C, CSSRS <sup>0</sup> , | | | х | | | x | | x | | |
| SRRS°, HAM-A° | 1 | | | | | | | | | |
| Self-Report Forms | | | X | | | X | | Х | | |
| Neurocognitive Tests | | | X | | | Х | | X | | |
| Computer Assessments | | | X | | | | | X | | |
| MRI Scan | - | | Х | | | Х | | X | | |
| Blood test_PT, PTT | 1 | | <del> </del> | | | | | [X] | F) (7 | |
| Lumbar Puncture (Optional) | | | l | | | | | | [X] | |

: Visit 2: Infusion: see below for abbreviations, \*\*Unless

Document Approved On: «ApproveDate»

\*Baseline will occur over 2 visits: Visit 1: MRS, blood and Symptom Domain Assessments; Visit 2: Infusion; see below for abbreviations, \*\*Unless prior documentation available from previous study, <sup>0</sup>Screening (or Baseline 1) and Week 2 only, [] indicates option to complete assessment, \*\*\* PCL-5 (with LEC) at Baseline 1 only, and PCL-5 (without LEC) at Day 3 and Week 2

## Types of Assessments will include:

- a. Psychiatric assessments
- b. Self report forms (to assess severity of depression, early life trauma)
- c. Neurocognitive testing
- d. Medical history and physical exam
- e. Blood sampling
- f. MRS scans-completed on 3 of your visits
- g. Lumbar puncture (optional)

**Screening Visit(s):** (Duration: approximately 7-8 hours and may be spread across more than one visit if needed).

Participation in this study requires a screening visit at which time your eligibility will be reviewed and verified. After you sign the consent form, a study clinican will ask you about your medical condition and mental health. The doctor or nurse practitioner will also conduct a physical examination. You will receive an electrocardiogram (EKG) to make sure you have no heart abnormalities and a chest x-ray to screen for tuberculosis. Approximately 5 teaspoons of your blood will be drawn to check for any abnormalities that would disqualify you for study participation. This includes testing for the human immunodeficiency virus (HIV), hepatitis B virus (HBV) and hepatitis C virus (HCV). You will be excluded from the study and referred to your primary care physician should you test positive for any of these viruses.

Your blood will also be evaluated for a marker of inflammation called C-reactive protein and other tests to assess your general medical status including tests to assess your blood, kidney, thyroid and liver status. You may have one or two drops of blood collected by trained research staff from a finger prick to measure inflammation level. You will also have a tuberculosis blood test. This test requires a small blood draw. If the test is positive for tuberculosis you will not be able to enter the study and the study doctor will recommend that you contact your primary care doctor for a referral to a TB specialist. You will be excluded from the study if you have TB and need INH treatment. You will also receive a pregnancy test if you are a female. You will be disqualified from the study if you are pregnant. If you are a woman of childbearing age we will ask you for documentation of adequate birth control during the study period. The screening process will take in total approximately 7-8 hours, but can be spread out over at least two visits if needed, and will occur either at the Emory Clinic Building B, 1365B Clifton Rd, or the Atlanta Clinical Translational Science Institute (ACTSI) in the Emory University Hospital. You are strongly encouraged to ask the study doctor or a member of the study staff if you have questions about the results of your lab tests and other diagnostic procedures.

If you qualify for the study and choose to enroll you will participate in 7-9 visits (including screening visits) across ~ 4 weeks. All study visits will take place either at Emory Clinic Building B or the Atlanta Clinical Translational Science Institute (ACTSI) outpatient research unit in the Emory University Hospital on the main Emory campus. At all visits you will fill out several self-report questionnaires that will ask about depressive symptoms and about the quality of your life. In terms of research, your blood will be looked at to see whether a decrease in depression following the infliximab infusion is associated with a decrease in inflammation chemicals. At each of these visits approximately eight teaspoons of your blood will be withdrawn to do routine laboratory checks and also for research purposes. Study visits will range in 4-8 hours of your time.

At screening and each visit, you will be asked to supply approximately 4 tablespoons of urine in a special cup that will test for the presence of drugs of abuse, such as marijuana, cocaine or heroin. A positive test for any of these drugs at screening will prevent you from participating in the study. A positive test at any other visits may


Document Approved On: «ApproveDate»

be a reason for withdrawing you from this study. Additionally, you will be asked to supply approximately 4 tablespoons of urine in a different cup that will be used to test for the presence of an infection.

Vital signs, including pulse and blood pressure, as well as weight will be measured at every visit. Height and waist circumference will be measured at screening. You may be asked to come in for additional screening visits to repeat any lab work or assessments.

## **Baseline Visits 1 & 2**

## **Baseline 1**: (Duration approximately 8.5 hours)

You will arrive to Emory Clinic Building B in the morning of your Baseline 1 visit. You will be asked to avoid Benadryl, alcohol, cigarettes, and foods high in MSG (for example, Chinese fast food, frozen dinners, or other processed foods) 24 hours prior to this visit. You will be asked not to eat or drink anything but water after midnight the night before your visit, planning for blood to be drawn first thing in the morning. You will be asked to give a small sample of blood, about 5 teaspoons collected from a vein in your arm by an Emory Healthcare professional, to measure your inflammation level and to look at your genes related to inflammation and metabolism. You will also give a urine sample in order to test for any signs of infection and drugs of abuse. After the blood draw, you will be able to eat and drink as normal until two hours before your scan, when you will be asked to not eat or drink anything but water. You will undergo a study medical evaluation with a doctor or nurse practitioner and will have your vital signs checked. You will be asked questions about how you are feeling and fill out questionnaires intended to measure the current level of emotional distress and other symptoms pertaining to mental health. The fasting research and safety lab tests, medical evaluation, and self-report behavioral assessments will take about 60-90 minutes.

You will then have a  $\sim$  30 minute break following which you will complete paper and pencil and computerized neuropsychological tests. You will complete a series of computer-based tests intended to measure your cognitive abilities including attention, concentration, memory and reaction time. You will also complete a series of computerized decision-making tasks that will require you to select different options using different buttons. These tasks measure your level of motivation. Some tasks will require you to make your responses very rapidly. On these tasks, you will have the opportunity to earn additional payment based on your task choices and performance. You will receive this payment by check in the mail. The assessments and tests will take about  $\sim$  90 minutes.

You will then be escorted to the scan room where you will undergo MRI scans for 2.5 hours (maximum). The MRS scan is being done to identify brain changes resulting from high inflammation in the body. You will be walked by study staff to the Emory University Imaging Facility and enter a large room where the MRI scanner is located. This scanner uses a very strong magnet to take pictures of your brain. MRI scans are painless and contain no radiation. You will be asked to remove all jewelry and other metal-containing objects. You will then be placed on a narrow table, which will slide into the MRI scanner. The scanner is a large closed box with a tube in the middle. You will lie in the tube while the scan is being done. The tube is about 6 feet long and 25 inches wide. You will then be asked to lie still during the scan for about 90 minutes.

As part of the scanning process, you will be fit with a head coil, which resembles a larger frame football helmet for the entire duration of the scanning period. You will be able to communicate with the scanning personnel using a microphone and speaker in the scanner bore. You will hear some loud noises as the scanner takes pictures of your head. You will be offered earplugs to wear while you are being scanned to decrease how loud the noise seems to you. Occasionally, people have an extreme fear reaction (claustrophobia) to being in the scanner. If this occurs you will be removed from the scanner and the experiment will be stopped. You will be given a short break (lasting for 15 minutes) an hour into the scan. After the scan you may eat and drink as normal. The scans will take approximately 120-150 minutes total. You will repeat the MRI scanning procedure on Visit Dav 3 and Week 2.

Your total time commitment for this visit will be approximately 8.5 hours with breaks.


If there is a considerable break between study visit procedures (i.e. a lapse of at least 2 hours outside of the total time commitment), you may leave and then return to complete the visit, and will be compensated an additional study visit's compensation.

Baseline 2 (Infusion): (Between 1-7 days after Baseline 1; duration approximately 4-5 hours)

You will be escorted to ACTSI-CRN where you will complete routine lab work checking for signs of infection. There you will be randomly assigned (similar to a flip of a coin) to receive either infliximab or placebo (an inactive compound). You have a one in two chance of receiving infliximab and a one in two chance of receiving placebo. If you receive infliximab, your dose will be 5 milligrams for every kilogram of your body weight. The placebo will be salt water. Neither you nor the study doctor will know whether you receive infliximab or placebo because all subjects will receive their infusions from identical appearing bags that have been specially prepared for the study. However, if a medical emergency occurs, the information about whether you received infliximab or placebo is available to your study doctor.

During the infusion visit, a study nurse or doctor will review your medical history with you and also complete a physical examination. A trained study staff member will complete a clinical interview with you and ask you about any bad reactions to a study procedure. Your height, weight, and vital signs will be recorded again at this visit. You will be asked to supply about 4 tablespoons of urine in a special cup. This will test for the presence of drugs of abuse, such as marijuana, cocaine or heroin. A positive test for any of these drugs at screening will prevent you from participating in the study. A positive test at any other visits may be a reason for withdrawing you from this study. Also, you will be asked to supply about 4 tablespoons of urine in a different cup that will be used to test for the presence of any infections or drugs of abuse.

For the infusion, you will sit in a special chair and a trained nurse will place an intravenous (IV) needle in a vein in your arm. Some of your blood will be drawn through the IV for routine labs and for research purposes before you receive the infusion, as described above. It will take about 2 hours for the infusion to be completed. You will be monitored for any type of bad reaction, such as an allergic response, during the infusion and for about 10-20 minutes afterwards. The nurse at the center where you receive the infusion or one of the nurses or doctors on the study team may ask you to stay longer if they think it is best for your safety. Your total time commitment will be approximately 4-5 hours.

Note: In some cases we will use a medicine similar to Infliximab in its place. This medicine, Inflectra, is an Infliximab biosimilar. This means that Inflectra is very similar to Infliximab but is not identical. While there may be some small differences between Inflectra and Infliximab, there are no clinically important differences in terms of safety and purity of the medicine. Inflectra is approved by the FDA for the same conditions as Infliximab. Please note each time you see Infliximab mentioned in this form, that Inflectra may be used instead.

## Post-Infusion Visits: Day 1, Day 3, Week 1, Week 2 (spread across 2 visits)

**Optional - Day 1 & Week 1:** (Duration approximately 2-3 hours)

Study visits Day 1 and Week 1 are optional. If you choose to participate in either one or both of the visits, you will come to the Emory Behavioral Immunology Program in the Emory Clinic, Building B in the morning. You will also be asked not to eat or drink anything but water the night before, in preparation for a fasting research blood sample draw. You will also give a urine sample in order to test for signs of infection and any drugs of abuse. You will undergo a short medical evaluation, in which a nurse practitioner or trained study staff member will take your vital signs, pulse, blood pressure, and weight, and ask you how you have been feeling since your infusion visit

Your total time commitment for each visit will be approximately 2-3 hours.

Day 3 & Week 2-Visit 1: (Duration approximately 7.5 hours)

Just like the Baseline 1 Visit, you will arrive to the Emory Behavioral Immunology Program in the Emory Clinic, Building B in the morning. You will be asked to avoid Benadryl, alcohol, cigarettes, and foods high in MSG (for example, Chinese fast food, frozen dinners, or other processed foods) 24 hours prior to these visits. You will also be asked not to eat or drink anything but water the night before, planning for blood to be drawn first thing in the morning. You will give a urine sample in order to test for signs of infection and any drugs of abuse. After the blood draw, you will be able to eat and drink as normal until two hours before your scan, when you will be asked to not eat or drink anything but water. You will undergo a short medical evaluation with a nurse practitioner or trained study staff member, who will take your vital signs and ask you how you have been feeling since your previous visit. You will be asked questions about how you are feeling and fill out questionnaires intended to measure the current of level of emotional distress and other symptoms pertaining to mental health. The study medical evaluation, fasting research and safety lab tests and self-report behavioral assessments will take ~ 60-90 minutes.

You will then have a  $\sim$  30 minute break following which you will complete the same paper and pencil neuropsychological tests you did at Baseline Visit 1, but only complete the computerized assessments at Week 2, Visit 1. You will receive payment for these tasks by check in the mail. The assessments and tests will take about  $\sim$  60-90 minutes.

You will then undergo MRI scans for 2.5 hours (maximum). You will be walked by study staff to the Emory University Imaging Facility and enter a large room where the MRI scanner is located. You will be asked to remove all jewelry and other metal-containing objects. You will then be placed on a narrow table, which will slide into the MRI scanner. You will be asked to lie still in the tube while the scan is being done for about 90 minutes. After the scan, you may eat and drink as normal. The scans will take approximately 120-150 minutes. Your total time commitment for each visit will be approximately 7.5 hours with breaks.

If there is a considerable break between study visit procedures (i.e. a lapse of at least 2 hours outside of the total time commitment), you may leave and then return to complete the visit, and will be compensated an additional study visit's compensation.

**Optional - Week 2-Visit 2 (Lumbar Puncture):** (Within 2 weeks of Week 2-Visit 1; Duration approximately 6 hours)

You may be asked to come in for an additional visit, which will consist of a lumbar puncture. This portion of the study is optional. If you choose to participate in this portion of the study, you will arrive at ACTSI-CRN (Research Unit inside Emory University Hospital). You will have a fasting research blood sample drawn following which you will be given a bag of saline through an IV in your arm. After 2-4 hours, you will have a spinal tap (Lumbar puncture or LP) in addition to the blood draw. The LP procedure allows us to collect a sample of your spinal fluid for the purpose of measuring inflammatory markers. An anesthesiologist from Emory University with considerable experience in performing spinal taps will conduct the procedure. Before the procedure, you will be offered pre-LP sedation with Versed through IV. The procedure will involve inserting a special long bore needle into the spine to obtain about 10ml (two teaspoons full) of fluid. This is a safe procedure and is often used to identify and treat brain diseases. It is possible that multiple attempts could be made to obtain the fluid. However, you have the ability to stop at any time. The procedure would be carried at a research unit dedicated to aid in such procedures by personnel who are well trained in conducting these procedures. Following the LP you will be instructed to rest till the research nurse determines that it is safe for discharge. You will be carefully observed for any side effects prior to discharge. A family member or friend will need to drive you home from the hospital after discharge. The nurse practitioner or designee will also make a follow-up call 1, 3, 7, and 14 days following the LP to check if you are experiencing any other study emergent side effects including chronic pain.

Your total time commitment will be approximately 6 hours.

**30-Day Phone Call** - Around one month after the infusion, you will receive a follow-up phone call from the coordinator or study staff member. He or she will ask you questions to make sure you have not had a bad reaction to anything that happened in the study.

 IRB Form 04152016

## Optional-Emory Department of Psychology 2-Visit (Functional MRI) fMRI Study

Study participants may choose to complete 2 additional study visits as an optional extension of this study. These visits are a part of a Task-Based Functional MRI (fMRI) study under the Department of Psychology, Dynamics of Inflammation and its Blockade on Motivational Circuitry in Depression, IRB#00087941 (see Table 1B). The purpose of the study is to see how the brain processes different types of information, and the way this affects behavior.

If you decide to participate, you will review and sign a separate consent form. If you complete the optional 2 visit study, you will be compensated approximately \$800 (in addition to the amount of compensation you receive for the main study). Both visits will take place on campus at the Emory Department of Psychology. At all visits, a study clinician will ask you questions about symptoms of depression using a standardized interview. You will also fill out several self-report questionnaires. These will ask about depressive symptoms and about the quality of your life. You will also be asked to complete some computer tasks and undergo a functional MRI scan which means you will be doing tasks while lying in the scanner. At each visit, they will collect a urine sample to test for drugs that may be present in your body and complete a pregnancy test if applicable.

Study Visit Schedule (including the optional 2-visits):

| Extra Visit 1 ** | Baseline | Infusion | 1-Day | 3-Day | 7-Day | 14-Day | Extra<br>Visit 2<br>** | LP |
|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|

## What are the possible risks and discomforts?

The most common risks and discomforts expected in this study are:

There may be risks, discomforts or side effects that are not yet known. The use of infliximab to treat major depression has not been approved by the Food and Drug Administration. There is no information regarding side effects or serious reactions to infliximab in medically healthy patients who are being treated for major depression. A number of side effects and more serious reactions to infliximab have been reported in patients receiving the medication for the treatment of rheumatoid arthritis or Crohn's disease. The Food and Drug Administration (FDA) issued a Black Box Warning for this medication because patients in treatment with this product are at increased risk of infections, including worsening of symptoms that may lead to hospitalization or death. Please read the list of possible side effects below.

From studies of infliximab, 10-50% of patients on infliximab had the following frequent negative health events: mild allergic reaction to the medication, stomach pain, nausea, diarrhea, heartburn, upper respiratory tract infections, sore throat sinusitis, coughing, runny nose, rash, fatigue, fever, headache, joint pain, back pain, urinary tract infection and hypertension.

The following negative health events were reported occasionally (in 1-10% of patients receiving infliximab): shortness of breath, itchy skin, chest pain, an abscess, insomnia, depression and oral thrush.

Rare negative health events occurring in less than 1% of patients receiving infliximab included severe immediate allergic reaction to the medication, delayed allergic response to the medication, serious bacterial infections,

tuberculosis, fungus infections and death. Most of these infections occurred in patients who were taking other medicines that suppress the immune system while they were taking infliximab. If you elect to enter this study you will be tested for tuberculosis using the blood test. If this test is positive, you will be excluded from study participation. At screening you will be asked if you have any symptoms of infection or if you have a history of any chronic or serious infections. If you do, you will be excluded from the study. Because taking infliximab could make you more vulnerable to getting a fungal infection we will take a small amount of blood at week 10 and sent it to Emory University Hospital lab to test for fungal infection. An increased risk of infection has been noted in patients taking drugs like infliximab who are also taking a drug called anakinra. If your doctor has prescribed anakinra for you, you will not be eligible for this study.

Symptoms of severe immediate allergic reaction to infliximab can include hives (red, raised, itchy patches of skin), difficulty breathing, chest pain, and high or low blood pressure. Symptoms of serious delayed reaction may include fever, rash, headache, and muscle or joint pain. If allergic symptoms occur during or immediately after the infusion you will be evaluated by a study physician who is expert at treating these symptoms. There is a standard procedure in place at the Infliximab Infusion Center for treating allergic reactions. If you develop symptoms of a delayed reaction at home, or if you develop any of the negative health events listed above, you should contact the study doctor immediately by calling the Emory Clinic operator (available 24 hours a day ) at 404-778-5000 and page Bobbi Woolwine, MSW at pager ID#15375. The study coordinator will give you an emergency information contact card to keep in your wallet.

Infliximab has been reported to worsen a condition called congestive heart disease and to lead to increased deaths in patients with this condition. You will be asked about any history of heart disease. In addition, you will receive an electrocardiogram (EKG) at the Mood and Anxiety Disorders Program offices or the Emory Clinic. This test examines whether your heart is functioning normally. To be enrolled in this study, you will need to have a normal EKG and no history of heart disease. No known risks are associated with the EKG screening test. However, it is possible the gel or tape, used in the procedure, may cause skin irritation at the site of the electrode(s).

Infliximab has been rarely associated with reductions in white and red blood cells, as well as platelets. There have been reports of death from these blood cell abnormalities in patients taking infliximab, however it has not been established that infliximab directly caused these abnormalities. You will have your blood cells examined prior to receiving the single infusion and repeated at each study visit after the infusion. If your white blood cells, platelets or red blood cells are abnormal prior to the infusion you will be excluded from the study. If you have a drop in any of your blood cells after the first infusion you will be assessed for medical follow-up when appropriate as determined by the study physician(s)

Infliximab has been associated in rare cases with a variety of central nervous system conditions, including inflammation of the nerves of the eye, seizures or a demyelinating condition that resembles multiple sclerosis. The study doctor will ask you about any history of central nervous system disorders, such as multiple sclerosis or seizures. If you have a history of a central nervous system illness such as multiple sclerosis, Guillain-Barre syndrome or seizures, or have tingling or numbness in any part of your body, you will be excluded from study participation.

You will be asked if you have ever had an allergic reaction from being around, or handling rodents. If you have had such an allergic reaction you will not be able to participate in this study. You will also be asked if you have ever had an allergic reaction to medicines made from mouse chemicals. These medicines include basiliximab (Simulect), daclizumab (Zenapax), gemtuzumab ozogamicin (Mylotarg), rituximab (Rituxan) and trastuzumab (Herceptin). These medications are used for cancer and to stop transplanted organs from being rejected from the body. If you have ever had an allergic reaction to any of these medications you will not be able to participate in this study.

Infliximab may increase the risk of developing an autoimmune condition such as systemic lupus erythematosis

or multiple sclerosis, but this has not been established. At screening you will be asked whether you have a history of any autoimmune related disorders, including lupus and multiple sclerosis, but also other conditions such as Crohn's disease, ulcerative colitis, rheumatoid arthritis, ankylosing spondilitis, scleroderma, thyroid or parathyroid disease or sarcoid. If you have a history of any autoimmune condition you will not be eligible for this study.

It is not known whether receiving infliximab would increase the risks involved in receiving a modified live virus vaccine. For this reason you will be asked about whether you have received a vaccine within four weeks prior to study entry or whether you are scheduled to receive a vaccine during the study or for a month afterwards. It is very important that you not receive any modified live virus vaccines for a month before the study, during the study and for at least one month after you have finished the study. You will be ineligible to participate in this study if you have or will receive a vaccine during this period. Examples of common modified live virus vaccines include vaccines for smallpox (vaccinia), measles, mumps, rubella (MMR), varicella (chicken pox and shingles), yellow fever, and the oral vaccines for: influenza (flu), typhoid, and polio vaccines. The injectable forms of influenza (flu), typhoid, and polio are killed (inactive) vaccines.

People who have been treated for rheumatoid arthritis or Crohn's disease for a long time tend to be more prone to a type of blood cancer called lymphoma. There have been some patients that while taking infliximab developed other types of cancer, but the number of people taking infliximab that developed cancer does not seem to be much different from what you would expect to see in people who are not taking infliximab. It is not known whether brief treatment with infliximab is a risk for cancer in medically healthy subjects, such as in this study. If you have ever had any type of cancer in the past, including skin cancer, you will not be eligible to participate in this study.

In addition to risks related to taking infliximab there are other risks associated with participating in this trial.

Blood Draws: Collecting blood from a vein in someone's arm is a standard medical procedure, although sometimes there may be some minor pain or bruising. Fainting and infection at the site of the blood draw are also known risks. Because we will be looking at biochemical information in your blood, there may also be other risks that we currently don't recognize or expect. Results that are considered important for your safety such as signs of infection, changes in blood glucose or electrolyte concentrations will be provided to you or your primary care provider, after obtaining a consent from you by obtaining your signature on the form for release of information. The research information that is learned from studies of your samples may be used scientifically and may be used by the sponsor in other research. The results of the analysis of your samples WILL NOT be made available to you or to your referring health care professional. A research lab, not by an Emory Healthcare lab, will do the testing. Some samples may be sent to other labs for additional analysis. The results of the biochemical analysis will not be recorded in your medical record, nor will they be provided to third parties. As for the blood drawing, standard sterile procedure for blood withdrawal will be used. In addition, the volume of blood withdrawn for this study will not exceed 200 ml (about 13 tablespoons).

<u>Chest X-Ray:</u> You will be exposed to radiation from x-rays. These procedures are not necessary for your medical care and will occur because you participate in this study. The estimated radiation dose that you will receive is equal to or less than the natural environmental radiation the average person receives in the United States annually. The principal risk associated with a radiation dose is the possibility of developing a radiation-induced cancer later in life. The risk for radiation-induced cancer from this study is negligible.

<u>Psychiatric Assessments:</u> The psychiatric assessments may involve detailed questioning regarding memories or feelings. Discussing mental symptoms may bring up emotions that distress some people. To minimize this, you will be able to discuss any disturbing memories or feelings you may experience with the study staff. Research personnel will be careful not to cause psychological distress during any part of the psychiatric assessment. There is a possible social risk involved if sensitive information related to previous mental health treatment is accidentally released. To guard against this risk, we will use a number and not your name to identify personal information. All documents will be kept in a locked area, and only the researchers will

Document Approved On: «ApproveDate»

have a key. The study has been designated as sensitivity study and the information will not be included in your regular Emory Healthcare Chart.

**Computer Testing:** There are no known risks for the tests of your thinking ability.

<u>MRI</u>: The MRI scanner contains a very strong magnet. Therefore, you may not be able to have the MRI if you have any type of metal implanted in your body, for example, any pacing device (such as a heart pacer), any metal in your eyes, or certain types of heart valves or brain aneurysm clips. Someone will ask you questions about this before you have the MRI. If you are a woman of childbearing potential, there may be unknown risks to the fetus. Therefore, you will not be allowed to participate in the study if you are pregnant.

Because the MRI is performed in an enclosed narrow space, some people may experience extreme fear, shortness of breath, rapid heartbeat or claustrophobia. If this happens to you, you may ask to stop the scan immediately. Metallic objects implanted in the body may move or heat due to force from the magnet in the scanner. Therefore, you will be carefully screened for any type of metal objects in your body prior to receiving the scan. If you have metal objects/implants in your body that are considered risky by Federal Government MRI safety guidelines, you will not receive the scan. No other known risks are associated with receiving the MRI/MRS scan.

Lumbar puncture: Some of the side effects of this procedure include bruising at the site of needle insertion, infection, bleeding and headache (post-LP headache). To reduce risks associated with receiving an LP, an experienced physician will conduct the procedure under standard sterile conditions. Subjects will receive two liters of normal saline prior to the procedure. This has been found to reduce the incidence of post-LP headache. Subjects will lie flat for two hours after the procedure and will be observed in the outpatient research unit for the emergence of any significant adverse effects until the research nurse deems it safe for you to be discharged. If subjects develop a headache they will be treated with pain medication or application of blood patch. Very rarely, some individuals develop neurological symptoms following the procedure, in which they would be evaluated by the Emory Emergency Room Physicians and treated accordingly. The Department of Anesthesiology at Emory University has 24 hour coverage of the ACTSI-CIN if more emergent side effects develop following LP. In addition, the entire procedure will be conducted in the Emory research unit at ACTSI-CIN, which has immediate access to EKG monitoring, cardiac resuscitation equipment and is located in close proximity to the Emory University Hospital Emergency room. You will be encouraged to call your study doctor right away if you have any of these side effects:

- you feel faint, or unsteady on your feet, when you stand up after you have been sitting or lying down
- you have lost power or sensation of one or both your lower limbs
- you have a headache that is not relieved by several doses of painkillers
- you feel confused
- your neck feels sore and stiff
- you develop nausea or vomiting

#### Risks with Pregnancy

The study medication (infliximab or placebo) may involve currently unforeseeable risks to pregnant women, the embryo or fetus, or to children of nursing women. If you are a woman who is pregnant, breast feeding, or planning to become pregnant within the period of the study, you must not participate in the study. In addition, all women of childbearing potential are required to undergo pregnancy testing before entering the study. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant.

All women of child bearing potential must use a medically acceptable contraceptive throughout the study. This includes oral (birth control pills), double-barrier method, injectable or implantable, or mechanical contraception; women whose sexual partners have had a vasectomy or have received or are using mechanical contraceptive devices. Condoms plus spermicide should be used in addition to other contraceptive methods to provide protection against sexually transmitted diseases and to provide additional protection against pregnancy. Men


IRB Form 04152016

who are participating in this research study need to understand the possible danger of taking a drug whose effects on the fetus are unknown.

If you miss a period or think you might be pregnant during the study, you must notify the investigator immediately so that you can be withdrawn from the study. If you become pregnant during the study or within 15 days after your last dose of study medication and your pregnancy is carried to term, the study doctor will ask to follow the course of the pregnancy and delivery, as well as the condition of the newborn.

For women of childbearing potential, if you (a) plan to become pregnant, (b) become pregnant, (c) think you may have become pregnant, or (d) plan to discontinue contraception, you are required to notify the study doctor immediately.

The study medication taken in this study may also have unknown risks.

## Will I benefit directly from the study?

This study is not designed to benefit you directly. Your depression may improve while you are in this study but it may not, and it may even get worse. This study is designed to learn more about how the study drug infliximab may decrease inflammation and treat symptoms of depression. The study results may be used to help others in the future.

## Will I be compensated for my time and effort?

Our preferred method of compensation will be the use of Clincards. All payments are made using a personal payment card. We issue this to you for free. The payment card is a prepaid debit card. It can be used exactly like a MasterCard. We load money onto your card electronically every time you need to be paid. The card scheme is run by Greenphire, an independent company specializing in payments for research studies and clinical trials. To issue your card, we need to give Greenphire some of your personal information. Banks and other financial institutions can access this information if they need to verify your identity when you use your card.

Emory University is required by law to report any payments we make to the IRS. Research payments in cash or cash equivalents that exceed \$600.00 per calendar year must be reported to the Internal Revenue Service (IRS) by the University. The level of reimbursement for this study is at a level that the potential exists for the federal tax reporting to the IRS for your participation in this study. To do this, Emory University Department of Finance needs to keep your Social Security Number on file. We are asking you to allow us to communicate your name, address, date of birth, research study name and Social Security Number to Greenphire and Emory University Department of Finance. If you want to receive e-mail or text alerts when payments are made to you, we will ask you to provide your e-mail or phone number as well. All of this information will be stored on computers owned by Greenphire. Greenphire will not have access to any other information collected during this study. Full instructions about using your card are included when we issue it. Please ask if you have any questions or concerns about the card scheme.

Each of your visits will be prorated according to the table below. An additional \$25 will be provided to cover travel expenses for participants that travel equal to or greater than 50 miles one way to Atlanta. Please let us know if you have any questions regarding the compensation schedule.

**Table 2: Compensation Schedule** 

| Visit | Total Amount | Amount put on Clincard immediately after visit | Amount put on Clincard at the end of study participation |
|---|---|---|---|
| Intake | \$25 | \$25 | |
| (Visit Total) | \$25 | | |

 IRB Form 04152016 Version Date: 10/23/2019

| | | T | |
|---|---|---|---|
| Screening | | | |
| Psychiatric evaluation,<br>history and physical, EKG,<br>chest x-ray and lab work | \$50* | \$50* | |
| (Visit Total) | \$50 | | |
| Baseline Visit 1 | | | |
| Medical and psychiatric<br>assessments, lab work<br>research blood,<br>neurocognitive tests, and<br>self-report surveys | \$50 | \$50 | |
| Computer Motivation Tasks<br>(depending on choice made<br>on the computer) | \$5-\$100 | | \$5-\$100 |
| Complete Scan | \$300 | | \$300 |
| Incomplete Scan | \$25** | \$25** | |
| Extended break<br>(Visit Total) | \$50***<br>\$80-\$500 | \$50*** | |
| Baseline Visit 2 | 400-4300 | | |
| Infusion (Infliximab or placebo) and all scheduled assessments | \$150 | \$50 | \$100 |
| (Visit Total) | \$150 | | |
| Post-Treatment<br>Day 1 (Optional) | | | |
| Medical assessment, lab<br>work, research blood | \$50 | \$50 | |
| (Visit Total) | \$50 | | |
| Post-Treatment<br>Day 3 | | | |
| Medical assessment, lab<br>work, research blood,<br>neurocognitive tests, and<br>self-report surveys | \$50 | \$50 | |
| Complete Scan | \$300 | | \$300 |
| Incomplete Scan | \$25** | \$25** | |
| Extended break | \$50*** | \$50*** | |
| (Visit Total) | \$75-\$400 | | |
| Post-Treatment<br>Week 1 (Optional) | | | |
| Medical assessment, lab work, research blood | \$50 | \$50 | |
| (Visit Total) | \$50 | | |
| Post-Treatment<br>Week 2 | | | |
| Medical assessment, lab<br>work research blood,<br>neurocognitive tests, and<br>self-report surveys | \$50 | \$50 | |
| Computer Motivation Tasks | \$5-\$100 | | \$5-\$100 |
| Complete Scan | \$300 | | \$300 |
| Incomplete Scan | \$25** | \$25** | |
| Extended break | \$50***<br>\$80-\$500 | \$50*** | |
| (Visit Total) | ψ00-ψ000 | | |
| Post-Treatment Week 2-Visit 2 (Optional) | | | |
| Spinal Tap (Lumbar<br>Puncture) | \$500 | | \$500 |
| (Visit Total) | \$500 | | |
| Total Study<br>Compensation | \$560-\$2225 | | |
| Department of<br>Psychology 2-Day<br>Study (Optional) | \$800 Maximum | | |

## Emory University IRB IRB use only

\*=Screening visit may be divided across 2 visits and paid \$25 per visit

\*\*= Unable to complete scan leading to termination from the study

\*\*\*=Subject can leave and return to complete visit if break is a minimum of 2 hours

Document Approved On: «ApproveDate»

## What are my other options?

If you decide not to enter this study, there is care available to you outside of this research study. The study clinician will discuss these options with you. You do not have to be in this study to be treated for depression.

Taking part in this study, however, may make you unable to participate in some other research studies, if they exclude people who have taken certain treatments. You should discuss this with the researchers if you have concerns. You may wish to research other study options at websites like clinicaltrials.gov and ResearchMatch.org.

## How will you protect my private information that you collect in this study?

Whenever possible, a study number, rather than your name, will be used on study records. Your name and other identifying information will not appear when we present or publish the study results.

Study records can be opened by court order.

## Certificate of Confidentiality

There is a Certificate of Confidentiality from the National Institutes of Health for this Study. The Certificate of Confidentiality helps us to keep others from learning that you participated in this study. Emory will rely on the Certificate of Confidentiality to refuse to give out study information that identifies you. For example, if Emory received a subpoena for study records, it would not give out information that identifies you.

The Certificate of Confidentiality does not stop you or someone else, like a member of your family, from giving out information about your participation in this study. For example, if you let your insurance company know that you are in this study, and you agree to give the insurance company research information, then the investigator cannot use the Certificate to withhold this information. This means you and your family also need to protect your own privacy.

The Certificate does not stop Emory from making the following disclosures about you:

- Giving state public health officials information about certain infectious diseases,
- Giving law officials information about abuse of a child, elderly person or disabled person.
- Giving out information to prevent harm to you or others.

Giving the study sponsor or funders information about the study, including information for an audit or evaluation.

## **Storing and Sharing your Information**

Your samples, genomic data and health information will be stored and shared with other researchers. The samples and information will be available for any research question, such as research to understand what causes certain diseases (for example heart disease, cancer, or psychiatric disorders), development of new scientific methods, or the study of where different groups of people may have come from. You will not be able to request destruction of these samples in this study.

How is my Genetic Information Protected? What are the Risks?


The Genetic Information Nondiscrimination Act (GINA) is a federal law that generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we
  get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this
  research when making a decision to hire, promote, or fire you or when setting the terms of your
  employment.

Be aware that GINA does <u>not</u> protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance, and does not apply to employers with less than 15 employees.

In addition to GINA, the State of Georgia has laws that prohibit insurers from using genetic testing information for any non-treatment purpose. However, like GINA, this state law protection has exclusions: life insurance policies, disability income policies, accidental death or dismemberment policies, medicare supplement policies, long-term care insurance policies, credit insurance policies, specified disease policies, hospital indemnity policies, blanket accident and sickness policies, franchise policies issued on an insurance policy written as a part of workers' compensation equivalent coverage, or other similar limited accident and sickness policies.

#### Privilege

In the State of Georgia, your genetic information has special legal protections called "privilege," which means that the information cannot be used as evidence in a court. By signing this form and allowing us to use and disclose your genetic information for the purposes described in this consent, you waive any privilege with regard to that genetic information, meaning that the information loses this legal protection.

#### **Medical Record**

If you have been an Emory Healthcare patient before, then you already have an Emory Healthcare medical record. If you have never been an Emory Healthcare patient, you do not have one. An Emory Healthcare medical record will be made for you if an Emory provider or facility gives you any services or procedures for this study.

We will take reasonable steps to keep copies of this form out of Emory Healthcare's medical records system. If we aren't successful in keeping these forms out, despite our efforts, we will take steps to remove them. If they cannot be removed, we will take steps to limit access to them.

Emory Healthcare may create study information about you that can help with your care. For example, the results of study tests or procedures. These study results will be put in your Emory Healthcare medical record. Anyone who has access to your medical records will be able to have access to all the study information placed there. The confidentiality of the study information in your medical record will be protected by laws like the HIPAA privacy rule. State and federal laws may not protect the research information from disclosure.

The results of some study tests and procedures will be used only for research purposes and will *not* be placed in your medical record. For this study, those items include: Cognitive testing results, self-report forms, clinician administered evaluations, History and Physical, MRI/MRS scans and biological samples (blood and CSF samples) collected for research purposes.

Tests and procedures done at non-Emory places may not become part of your Emory medical record. Also, if you decide to be in this study, it is up to you to let your other health providers know.

 IRB Form 04152016 Version Date: 10/23/2019

Study No.: IRB00090667 Emory

Emory University IRB IRB use only

## In Case of Injury

If you get ill or injured from being in the study, Emory will help you get medical treatment. Emory and the sponsor have not, however, set aside any money to pay you or to pay for this medical treatment. The only exception is if it is proven that your injury or illness is directly caused by the negligence of an Emory or sponsor employee. "Negligence" is the failure to follow a standard duty of care.

If you become ill or injured from being in this study, your insurer will be billed for your treatment costs. If you do not have insurance, or if your insurer does not pay, then you will have to pay these costs.

If you believe you have become ill or injured from this research, you should contact telephone number. You should also let any health care provider who treats you know that you are in a research study.

## **Costs**

There will be no costs to you for participating in this study, other than basic expenses like transportation. You will not be charged for any of the research activities. If the study procedures result in any medical complications that would not fall under "injury" as discussed above, the cost of treatment for those complications may be charged to you or your insurance.

## Withdrawal from the Study

You have the right to leave a study at any time without penalty.

For your safety, however, you should consider the study doctor's advice about how to go off the study treatment. If you leave the study before the final planned study visit, the researchers may ask you to have some of the final steps done.

The researchers also have the right to stop your participation in this study without your consent for any reason, especially if they believe it is in your best interest or if you were to object to any future changes that may be made in the study plan.

## 30 Day Off-Study Policy

There may be situations based on your schedule or ours that require more than 30 days to occur between study visits. If this is the case, for the purposes of your care and safety, a research assistant will inform you of the delay and temporarily remove you from the study. In the meantime, you should feel free to start or resume any form of treatment. When you return for your next study visit, you will be reevaluated for study eligibility and re-consented by a study clinician or coordinator. Based on your status, we will continue the study where you left off and will use as much previously collected data as possible. However you may be asked to repeat some bloodwork or assessments to evaluate any changes in your status.

## **Authorization to Use and Disclose Protected Health Information**

The privacy of your health information is important to us. We call your health information that identifies you, your "protected health information" or "PHI." To protect your PHI, we will follow federal and state privacy laws, including the Health Insurance Portability and Accountability Act and regulations (HIPAA). We refer to all of these laws as the "Privacy Rules." Here we let you know how we will use and disclose your PHI for the main study and for any optional studies in which you may choose to participate.

## **Main Study**

PHI that Will be Used/Disclosed:

 IRB Form 04152016 Version Date: 10/23/2019

Document Approved On: «ApproveDate»

Document Approved On: «ApproveDate»


The PHI that we will use or share for the main research study includes:

- Medical information about you including your medical history and present/past medications.
- Results of exams, procedures and tests you have before and during the study.
- Laboratory test results.

## Purposes for Which Your PHI Will be Used/Disclosed:

We will use and share your PHI for the conduct and oversight of the research study. We will use and share your PHI to provide you with study related treatment and for payment for such treatment. We will also use and share your PHI to conduct normal business operations. We may share your PHI with other people and places that help us conduct or carry out the study, such as laboratories, data management centers, data monitors, contract research organizations, Institutional Review Boards (IRBs) and other study sites. If you leave the study, we may use your PHI to determine your health, vital status or contact information. We will use and disclose your PHI for the administration and payment of any costs relating to subject injury from the study

## Use and Disclosure of Your Information That is Required by Law:

We will use and disclose your PHI when we are required to do so by law. This includes laws that require us to report child abuse or abuse of elderly or disabled adults. We will also comply with legal requests or orders that require us to disclose your PHI.

## Authorization to Use PHI is Required to Participate:

By signing this form, you give us permission to use and share your PHI as described in this document. You do not have to sign this form to authorize the use and disclosure of your PHI. If you do not sign this form, then you may not participate in the research study or receive research-related treatment. You may still receive non-research related treatment.

## People Who will Use/Disclose Your PHI:

The following people and groups will use and disclose your PHI in connection with the research study:

- The Principal Investigator and the research staff will use and disclose your PHI to conduct the study and give you study related treatment.
- Emory may use and disclose your PHI to get payment for study related treatment and to run normal business operations.
- The Principal Investigator and research staff will share your PHI with other people and groups to help conduct the study or to provide oversight for the study.
- National Institute of Mental Health (NIMH) is the Sponsor of the study. The Sponsor may use
  and disclose your PHI to make sure the research is done correctly and to collect and analyze
  the results of the research. The Sponsor may disclose your PHI to other people and groups like
  study monitors to help conduct the study or to provide oversight for the study.
- The research team and the Sponsor may use and disclose your PHI, including disclosure to insurance carriers to administer payment for subject injury.
- The following people and groups will use your PHI to make sure the research is done correctly and safely:
  - Emory offices that are part of the Human Research Participant Protection Program and those that are involved in study administration and billing. These include the Emory IRB, the Emory Research and Healthcare Compliance Offices, and the Emory Office for Clinical Research.
  - Government agencies that regulate the research including: Office for Human Research Protections; Food and Drug Administration.
  - Public health agencies.
  - Research monitors and reviewer.

Accreditation agencies.

Sometimes a Principal Investigator or other researcher moves to a different institution. If this
happens, your PHI may be shared with that new institution and their oversight offices. PHI will
be shared securely and under a legal agreement to ensure it continues to be used under the
terms of this consent and HIPAA authorization.

## **Expiration of Your Authorization**

Your PHI will be used until this research study ends.

## **Revoking Your Authorization**

If you sign this form, at any time later you may revoke (take back) your permission to use your information. If you want to do this, you must contact the study team at:

At that point, the researchers would not collect any more of your PHI. But they may use or disclose the information you already gave them so they can follow the law, protect your safety, or make sure that the study was done properly, and the data is correct. If you revoke your authorization you will not be able to stay in the main study.

## Other Items You Should Know about Your Privacy

Not all people and entities are covered by the Privacy Rules. HIPAA only applies to health care providers, health care payers, and health care clearinghouses. If we disclose your information to people who are not covered by the Privacy Rules, including HIPAA, then your information won't be protected by the Privacy Rules. People who do not have to follow the Privacy rules can use or disclose your information with others without your permission if they are allowed to do so by the laws that cover them. The Sponsor, and people and companies working with the Sponsor on this study are not covered by the Privacy Rules. They will only use and disclose your information as described in this Consent and Authorization.

To maintain the integrity of this research study, you generally will not have access to your PHI related to this research until the study is complete. When the study ends, and at your request, you generally will have access to your PHI that we maintain in a designated record set. A designated record set is data that includes medical information or billing records that your health care providers use to make decisions about you. If it is necessary for your health care, your health information will be provided to your doctor.

We may remove identifying information from your PHI. Once we do this, the remaining information will not be subject to the Privacy Rules. Information without identifiers may be used or disclosed with other people or organizations for purposes besides this study.

If you decide to sign consent for enrollment into this study, there are a couple of items that you may opt to check on the signature pages. You do not have to check these items in order to be in the study. They are optional. The first item is whether or not you are willing to participate in the lumbar puncture procedure. If you are not willing to participate in the lumbar puncture procedure you may still participate in the study. The second item is agreeing to allow the results of your screening assessments and any data collected from you during the study to be shared with other research studies of your choosing. If you decide not to check this item you may still participate in the study.

 IRB Form 04152016 Version Date: 10/23/2019

Document Approved On: «ApproveDate»

Emory University IRB IRB use only

## **Contact Information**

Study No.: IRB00090667

Contact

- if you have any questions about this study or your part in it,
- if you feel you have had a research-related injury or a bad reaction to the study drug, or
- if you have questions, concerns or complaints about the research

Contact the Emory Institutional Review Board at 404-712-0720 or 877-503-9797 or irb@emory.edu:

- if you have questions about your rights as a research participant.
- if you have questions, concerns or complaints about the research.
- You may also let the IRB know about your experience as a research participant through our Research Participant Survey at <a href="http://www.surveymonkey.com/s/6ZDMW75">http://www.surveymonkey.com/s/6ZDMW75</a>.

Document Approved On: «ApproveDate»

## Consent and Authorization

## You are also free to agree or disagree to the option below:

In the box below, please put your initials under "Yes" if you agree to the statement, or "No" if you do not agree and then sign on the appropriate line below:

| Yes | No | |
|---|---|---|
| | | I DO agree to abstain from sexual intercourse 14 days prior to study infusion and to use a medically approved birth control method for the |
| | | duration of the study. If I am a woman, I HAVE been advised to delay conception for 6 months post-infusion. |
| <u>Yes</u> | <u>No</u> | LAM willing to participate in the LD precedure as described as page 9 of |
| | | I AM willing to participate in the LP procedure, as described on page 8 of this consent form. |
| Yes | No | LAM interested in month in the CAVIII Obode with the Foreign |
| | | I AM interested in participating in the 2-Visit Study with the Emory Department of Psychology, IRB#87941, as an optional extension of this study. |
| Yes | No | I DO agree, if I consent to participate in any additional studies, that the results of my screening tests (laboratory, medical, and psychiatric) and any data collected during my study visits for this project may be shared with the |
| | | study team of the project for which I gave consent. I also authorize the use of my PHI for this purpose. |
| Yes | No | May we contact you in the future regarding participation in future research |
| | | studies? You may then decide if you are willing to participate. |

## TO BE FILLED OUT BY SUBJECT ONLY

Please **print** your name, **sign**, and **date** below if you agree to be in the main study. By signing this consent and authorization form, you will not give up any of your legal rights. We will give you a copy of the signed form to keep.


| Study No.: IRB00090667 Name of Subject | Emory University IRB IRB use only | Docume | nt Approved On: «ApproveDate | |
|---|---|---|---|---|
| Signature of Subject (18 or | older and able to consent) | Date | Time | |
| | TO BE FILLED OUT BY STUDY TEAM | M ONLY | | = |
| Name of Person Conducting | g Informed Consent Discussion | <u> </u> | | |
| Signature of Person Condu | cting Informed Consent Discussion | Date | Time | |

 IRB Form 04152016
